CLINICAL TRIAL: NCT00844779
Title: Evaluation of Non Alcoholic Metabolic Liver Diseases in Patients Harboring Central Adiposity and Insulin Resistance by Biochemical and Functional Genomic Approaches
Brief Title: Molecular Investigation of Non Alcoholic Fatty Liver Diseases in Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Other Study IDs: 3966
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Liver Disease
Keywords: Metabolic syndrome- hepatic steatosis- steatohepatitis - gene expression; Non alcoholic fatty liver disease (NFALD)
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery; Cholecystectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- T: (n=30): without central adiposity, without insulin resistance, operated for cholecystectomy or a benign liver tumor.
  Interventions: Procedure: cholecystectomy or benign liver tumor removal
- A: (n=30): with central adiposity, insulin resistance and hepatic steatosis (histology).
  Interventions: Procedure: Bariatric surgery
- B: (n=30): with central adiposity, insulin resistance and steatohepatitis ± hepatic fibrosis (histology).
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Gastric bypass.
  Groups: A; B
Procedure: cholecystectomy or benign liver tumor removal — cholecystectomy or benign liver tumor removal
  Groups: T

SUMMARY:
Non alcoholic fatty liver diseases (NAFLD) are represented by two main pathological conditions, hepatic steatosis (HS) and non alcoholic steatohepatitis (NASH), which are characterized by the accumulation of fat in the liver. The diagnosis of these two entities is achieved by histology and neither imaging nor biochemical markers are accurate enough to discriminate them. At the contrary of HS, NASH features hepatocyte necrosis, inflammation and fibrosis of variable intensity that could progress and ultimately evolve to cirrhosis. Therefore, it is important to distinguish between HS and NASH in order to treat the patients accordingly. In this study, the investigators aim to understand the molecular mechanisms that govern the transition from benign steatosis to complicated NASH. The investigators will analyze by "Q-RT-PCR" and "DNA microarray" technologies in the liver of obese patients, the expression of genes that are susceptible to be involved in the pathogenesis of NAFLD and identify the potential signaling pathways responsible for the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Group T(n=30): patient without central adiposity, without insulin resistance, operated for cholecystectomy or a benign liver tumor
* Group A (n=30): patient with central adiposity, insulin resistance and hepatic steatosis (histology).
* Group B (n=30): patient with central adiposity, insulin resistance and steatohepatitis ± hepatic fibrosis (histology).

Exclusion Criteria:

* viral or autoimmune hepatitis
* hematochromatosis
* alcohol consumption (> 20 g/24h women, >30 g/24h men)
* type 1 diabetes
* inflammation or infection before procedure
* abnormal hemostasis or coagulation- pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michel DOFFOEL, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Service d'Hépato-Gastro-Entérologie - Nouvel Hôpital Civil, Strasbourg
  - Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil, Strasbourg